CLINICAL TRIAL: NCT00295334
Title: Moderate Alcohol Intake Among Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iris Shai (Other)
Collaborators: The Israeli Diabetes Research Group (Unknown); Hadassah Medical Organization (Other); Soroka University Medical Center (Other); Julio Vainstein, Wolfson Medical Center, Holon, Israel (Unknown); Tishbi Wines, Israel and Admiral Wine Imports, US (Unknown); Harvard University (Other)
Responsible Party: Sponsor-Investigator, Iris Shai, Prof., The S. Daniel Abraham International Center for Health and Nutrition
Organization: The S. Daniel Abraham International Center for Health and Nutrition (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 250505
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: adherence; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ethanol

ARMS (3):
- Mediterranean diet + red wine (Active Comparator)
  Interventions: Drug: alcohol
- Mediterranean diet + white wine (Active Comparator)
  Interventions: Drug: alcohol
- Mediterranean diet+ mineral water (Placebo Comparator)
  Interventions: Drug: alcohol

INTERVENTIONS:
Drug: alcohol

SUMMARY:
Our specific aim is to explore the effect of moderate alcohol intake on parameters of glycemic index and lipid profile among patients with type 2 diabetes.

DETAILED DESCRIPTION:
Successful long-term control of hyperglycemia decreases the risk for diabetic complications . Although a family history of diabetes is an established risk factor for type 2 diabetes, lifestyle factors also play an important role in its cause . However, physicians are poorly informed about how their patients' alcohol use affects risk for or management of diabetes. Moderate alcohol consumption has been associated with lower risk of both cardiovascular disease and type 2 diabetes, and is also linked to lower cardiovascular risk among type 2 diabetics. Potential mechanisms have focused primarily on lipid metabolism, coagulation, fibrinolysis, and insulin sensitivity. A recent systematic review of the literature to assess the effect of alcohol consumption on risk for and management and complications of diabetes mellitus suggests that moderate alcohol consumption is associated with a decreased risk for diabetes, whereas heavy alcohol consumption may be associated with an increased risk. Our aim is to assess the effect of moderate alcohol intake on glycemic control and cardiovascular disease mediators among patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-75 yrs.
2. Alcohol abstainers (less than or equal to 1 drink/week)
3. Established diagnosis of type 2 diabetes.
4. Clinically stable, with no stroke or MI within the last 3 months and no major surgery within the last 3 months.

Exclusion Criteria:

1. Taking Insulin >2 injections /day, or with insulin pump.
2. TGs>500 mg/dL.
3. HbA1c >10%
4. Serum creatinine > 2 mg/dl
5. Liver dysfunction (above 2 fold level of ALT and/or AST enzymes)

5. Evidence of severe diabetes complications (such as proliferative retinopathy or renal disease).

6. Patients with autonomic neuropathy manifested as postural hypertension and/or hypoglycemia unawareness. 7. Using drugs that might significantly interact with moderate alcohol. List of drugs will be obtained from pharmacology expert. 8. Presence of active cancer, receiving or had received chemotherapy in last 3 years.

9. Suffering a major illness that might probably require hospitalization (upon physician's evaluation).

10. Clinically assessed as having high potential of addictive behavior as judged by a validated clinical assessment and/or personal or family history of addiction, alcoholism or alcohol abuse.

11. Severe symptoms during run-in as assessed by the physician. 12. Pregnant or lactating women. 13. Participation in another trial in which active intervention is being received.

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Shai, RD PhD, Principal Investigator — Ben-Gurion University of the Negev

REFERENCES:
- [Derived] Shai I, Wainstein J, Harman-Boehm I, Raz I, Fraser D, Rudich A, Stampfer MJ. Glycemic effects of moderate alcohol intake among patients with type 2 diabetes: a multicenter, randomized, clinical intervention trial. Diabetes Care. 2007 Dec;30(12):3011-6. doi: 10.2337/dc07-1103. Epub 2007 Sep 11. PMID 17848609
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/17848609/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: All participants received individual dietary counseling by registered dietitians trained to work with type 2 diabetic patients. Each dietitian reinforced identical nutritional strategies to achieve glycemic control in both study groups but did not specifically try to promote weight loss. Reinforcement of dietary counseling for both groups was based on the American Diabetes Association recommendations for patients with type 2 diabetes, which include 45-60% calories from carbohydrates, up to 30% from fat (with restriction of saturated fat to <7% of total calories and minimization of trans fat), and 15-20% from protein.
  Participants randomly assigned to the control group were instructed to drink 150 ml of the nonalcoholic diet malt beer we provided, using the same standard measured glass, during dinner.
- Alcohol: All participants received individual dietary counseling by registered dietitians trained to work with type 2 diabetic patients. Each dietitian reinforced identical nutritional strategies to achieve glycemic control in both study groups but did not specifically try to promote weight loss. Reinforcement of dietary counseling for both groups was based on the American Diabetes Association recommendations for patients with type 2 diabetes, which include 45-60% calories from carbohydrates, up to 30% from fat (with restriction of saturated fat to <7% of total calories and minimization of trans fat), and 15-20% from protein.
  the alcohol group was instructed to reduce carbohydrates by 100 kcal, but not at dinner, to decrease the likelihood of alcohol-induced hypoglycemia.
  Patients assigned to consume alcohol were instructed to start drinking gradually (over a 2-week period) 150 ml of wine (13% alcohol, 13 g) that we provided, using a standard measured glass, during dinner. The patients could choose either dry red (Merlot) or white (Sauvignon Blanc) wine.
Period: Overall Study
Arm/Group | Control | Alcohol
Started | 34 | 75
Chosen Wine (Red, n) | 0 | 56
Completed | 25 | 66
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Alcohol: All participants received individual dietary counseling by registered dietitians trained to work with type 2 diabetic patients. Each dietitian reinforced identical nutritional strategies to achieve glycemic control in both study groups but did not specifically try to promote weight loss. Reinforcement of dietary counseling for both groups was based on the American Diabetes Association recommendations for patients with type 2 diabetes, which include 45-60% calories from carbohydrates, up to 30% from fat (with restriction of saturated fat to <7% of total calories and minimization of trans fat), and 15-20% from protein.
  the alcohol group was instructed to reduce carbohydrates by 100 kcal, but not at dinner, to decrease the likelihood of alcohol-induced hypoglycemia.
  Patients assigned to consume alcohol were instructed to start drinking gradually (over a 2-week period) 150 ml of wine (13% alcohol, 13 g) that we provided, using a standard measured glass, during dinner. The patients could choose either dry red (Merlot) or white (Sauvignon Blanc) wine; 75% chose red wine.
- Total: Total of all reporting groups
Arm/Group | Alcohol | Control | Total
Number analyzed (Participants) | 75 | 34 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (6.9) | 61.1 (6.7) | 61.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 13 | 46
  Male | 42 | 21 | 63
Region of Enrollment [Number; unit: participants]
  Israel | 75 | 34 | 109

OUTCOME MEASURES:

1. Primary Outcome: Glucose
Description: A change from baseline to 3-month time points is reported
Time Frame: Differance between 3 month time point minus baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alcohol | Control
Number analyzed (Participants) | 75 | 34
mg/dL | -21.55 (41.18) | 1.92 (25.69)

2. Primary Outcome: Adherence
Description: Count of participants that finished the 3-month intervention
Time Frame: Adherence at 3-months (end of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol | Control
Number analyzed (Participants) | 75 | 34
Participants | 66 | 25

3. Primary Outcome: HbA1c
Description: A change from baseline to 3-month time points is reported
Time Frame: Differance between 3 month time point minus baseline
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Alcohol | Control
Number analyzed (Participants) | 75 | 34
% of HbA1c | -0.29 (0.99) | -0.24 (0.86)

4. Secondary Outcome: LDL, HDL, TG
Description: Differance between 3 month time point minus baseline
Time Frame: A change from baseline to 3-month time points is reported
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Alcohol | Control
Number analyzed (Participants) | 75 | 34
mg/dl
  LDL | -11.53 (29.22) | 0.12 (24.03)
  HDL | -2.34 (9.85) | -3.0 (4.55)
  TG | 23.05 (81.10) | 10.40 (87.86)

ADVERSE EVENTS:
Arm/Group | Alcohol | Control
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/34
Other Adverse Events (participants affected / at risk) | 3/75 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alcohol (N=75) | Control (N=34)
gastric pain (Gastrointestinal disorders) | 1 | 0
illness (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No